CLINICAL TRIAL: NCT07114250
Title: Comparative Study Between Spinal Anesthesia Versus General Anesthesia in Patients Undergoing Supine Percutaneous Nephrolithotomy
Brief Title: Comparative Study Between Spinal Anesthesia Versus General Anesthesia in Supine Percutaneous Nephrolithotomy Operation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Mahmoud Ibrahim Hamouda, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36264MS737/11/24
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-05

CONDITIONS: Spinal Anesthesia; Percutaneous Nephrolithotomy; General Anesthesia
Keywords: General Anesthesia; Percutaneous nephrolithotomy; Spinal Anesthesia; Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Anesthesia (Experimental): Spinal Anesthesia: Patients included in this group will undergo supine Percutaneous nephrolithotomy under spinal anesthesia
  Interventions: Procedure: spinal anesthesia
- General Anesthesia (Experimental): Patients included in this group will undergo supine Percutaneous nephrolithotomy under general anesthesia.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Spinal Anesthesia group: Patients included in this group will undergo supine Percutaneous nephrolithotomy under spinal anesthesia
  Arms: Spinal Anesthesia
Procedure: General Anesthesia — General Anesthesia : Patients included in this group will undergo supine Percutaneous nephrolithotomy under general anesthesia
  Arms: General Anesthesia

SUMMARY:
The aim of this study is to evaluate the efficacy of spinal anesthesia as an alternative to general anesthesia in PCNL operation in supine position.

DETAILED DESCRIPTION:
Nephrolithiasis remains a common health problem around the globe. Percutaneous nephrolithotomy is the preferred modality for large and complex renal calculi. Percutaneous nephrolithotomy is the treatment of choice for calculi which fail treatment with extracorporeal shockwave lithotripsy and ureteral endoscopy.

There are variations to Percutaneous nephrolithotomy, including position, imaging modality, dilatation method, and anesthesia method. There is conflicting evidence between the appropriate use of general anesthesia versus spinal anesthesia for Percutaneous nephrolithotomy

The conventional position of Percutaneous nephrolithotomy is prone, which allows direct access to the posterior calyx with minimal risk of bowel puncture.

However, this positioning method limits the possibility of switching anesthesia from regional to general. The alternative position is supine Advantage in this position is that the spine does not overlap with kidney and fluoroscopic visualization can be achieved.

Nowadays, Percutaneous nephrolithotomy is usually performed under general anesthesia from a urological perspective, the particular advantages of general anesthesia in Percutaneous nephrolithotomy procedure include its feasibility to control tidal volume, secure patient airway, and extensibility of anesthesia time. The feasibility of controlling tidal volume minimizes renal mobility secondary to respiration while the extensibility of anesthesia time allows the surgeon to create multiple punctures with subsequently increased efficacy of the procedure . Despite the superior results of Percutaneous nephrolithotomy surgeries under general anesthesia, it has found to be associated with certain disadvantages such as its high cost and higher incidences of drug interactions. The incidence of complications is high especially when the position of patient is changed from supine to prone position. Common complications associated with use of general anesthesia i.e. injury to lung, brachial plexus, tongue and occasionally to spinal cord are its major drawback. Other minor but common side effects include postoperative nausea and vomiting On the other hand, there are recent reports regarding the use of spinal anesthesia in Percutaneous nephrolithotomy demonstrating lower post-operation pain, less drug intake, less bleeding, and reduces venous pressure in the surgery field .A limited number of prospective randomized trials have been carried out to establish which one of these procedures is better at decreasing perioperative complications. The influence of the type of anesthesia on the effectiveness of Percutaneous nephrolithotomy remains uncertain. Thus, the aim of this study is to evaluate the efficacy of spinal anesthesia as an alternative to general anesthesia in Percutaneous nephrolithotomy operation in supine position.

The aim of this study is to evaluate the efficacy of spinal anesthesia as an alternative to general anesthesia in Percutaneous nephrolithotomy operation in supine position.

Primary outcome:

• Patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years old.
* Both sexes.
* American Society of Anesthesiologists physical status (I- II).
* Patient with single renal stone size 2-3cm prepared for supine Percutaneous nephrolithotomy

Exclusion Criteria:

* Patient refusal.
* Pregnancy
* Morbid obese with Body mass index > 35 kg/m2.
* Contraindication for spinal anesthesia.
* Renal anomalies (horseshoe kidney, ectopic kidney).
* Presence of multiple stones or staghorn stones.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-05-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 24 hours
  Degree of patient satisfaction will be assessed according to a 5-point Likert scale (5: excellent, 4: Good, 3: Satisfactory, 2: Poor, 1: Very poor)

SECONDARY OUTCOMES:
Visual analog scale | 24 hours
  Visual analog scale will be assessed after surgery over 24 hours using as (0 = no pain and 10 = intolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Aya Hamouda, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF